CLINICAL TRIAL: NCT04110678
Title: Nasal Administration of the NeuroEPO in Parkinson Disease: Short-term Tolerance Physician Lead Trial
Brief Title: Tolerance to NeuroEPO in Parkinson Disease
Acronym: NeuroEPO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Center for Neurological Restoration, Cuba (Other)
Collaborators: Center of Molecular Immunology, Cuba (Other); University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Ivonne Pedroso Ibanez, Head of Movement Disorders Clinic, International Center for Neurological Restoration, Cuba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NeuroEPO-001-PD
Record Dates: First submitted 2019-09-18; First posted 2019-10-01 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Tolerance; NeuroEPO; side effects; UPDRS; Cognition
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, Physician lead trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be performed by the promoter institution Centro Inmunologia Molecular from Spanish CIM who assigned the selected patients to two groups neuroEPO and placebo giving a code. The specialists at CIREN didn't have access to the information. Both groups received a vial of the molecule with identical organoleptic characteristics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeuroEPO (Active Comparator): The dose of NeuroEPO was a vial with a dose of 1 mL/1mg administered intra-nasally for five consecutive weeks.
  Interventions: Drug: NeuroEPO
- Placebo (Placebo Comparator): The dose of placebo was a vial with a dose of 1 mL/1mg of an intranasal inert solution administered intra-nasally for five consecutive weeks.
  Interventions: Drug: NeuroEPO

INTERVENTIONS:
Drug: NeuroEPO — NeuroEPO [CIMAB S.A, Havana, Cuba]
  Other Names: Placebo

SUMMARY:
Treatment strategies in Parkinson's disease (PD) can improve a patient's quality of life but cannot stop the progression of PD. The investigators are looking for different alternatives that modify the natural course of the disease and recent research has demonstrated the neuroprotective properties of erythropoietin. In Cuba, the Center for Molecular Immunology (CIM) is a cutting edge scientific center where the recombinant form (EPOrh) and recombinant human erythropoietin with low sialic acid (NeuroEPO) are produced.

DETAILED DESCRIPTION:
Delivery of therapeutic agents as erythropoietin (EPO) into Central Nervous System through intranasal route could benefit patients with neurological disorders. A new nasal formulation containing a non-hematopoietic recombinant EPO (NeuroEPO) has shown neuroprotective actions in preclinical models and the safety trial of NeuroEPO was evaluated for the first time in humans in Cuba.

The researchers previously conducted a proof of concept clinical trial, administering EPOrh subcutaneously where the neuropsychological performance was measured as a secondary endpoint. This protocol has the register number NCT01010802. Results showed an increased neuropsychological performance of patients after administration as compared to before administration results.

In this protocol two institutions were leading a physician clinical trial.The two institutions: International Center for Neurological Restoration (CIREN from Centro Internacional de Restauracion Neurologica from Spanish) where the recruitment and clinical evaluation of the PD patients will be done and the Center for Molecular Immunology, who was the promoter.

Randomisation will be performed by the CIM to assign the patients to groups. The groups will receive neuroEPO or placebo with identical organoleptic characteristics. The informed consent of all patients will be obtained before the start of the trial after the selection and primary evaluation of the inclusion criteria.

The dose of neuroEPO will be a vial with a dose of 1 mL/1mg administered intra-nasally for five consecutive weeks. The placebo group was administered 1 mL of an intranasal inert solution for the same period of time.

The IBM SPSS Statistics V 21 package will be used for the statistical analysis of the data. The investigators will use tables of frequency analysis and descriptive statistics to analyse the demographic characteristics of the sample.

The analysis of the results obtained will be done studying the differences between quantitative variables for paired and unpaired samples, the Wilcoxon and U of Mann-Whitney tests will be used respectively. For the qualitative variables Chi square (X2) test will be used. All values of p < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patient who fulfilled the London Brain Bank's operational criteria for PD
* Willing to participate in the study;
* ≥1 year since disease onset;
* Good response to antiparkinsonian treatment with levodopa (>30% change in motor score on the motor section of the Unified Parkinson's Disease
* no prior poly globulin (hematocrit ≤50%);

Exclusion Criteria:

* Refusal to participate;
* Known hypersensitivity to products derived from eukaryotes or hypersensitivity to human albumin;
* Pregnancy or breastfeeding;
* Hypertension;
* Immunosuppressant, androgen or anabolic steroid treatment in the month prior to recruitment;
* Sepsis or active infection;
* Active acute or chronic inflammatory diseases;
* Haematological diseases, such as sickle cell disease, myelodysplastic syndromes, active clotting or bleeding disorders;
* Malignant tumor or cancer treatment;
* Alcoholism or drug addiction in the two years prior to inclusion assessment.
* Significant cognitive decline as measured by clinical assessment, DRS (Dementia Rating Scale) and the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with local nasal events | day 1-5
  the administration of the drug is intra-nasal for that reason the first adverse event to study is the irritation of the nose. The presence of toxicity signs in the nasal mucous, such as: redness, swelling and nasal congestion was evaluated by means of thorough medical examination of the nasal cavity by the same Otorhinolaryngology Specialist.
Number or participants with increment in the haematological and biochemistry parameters | day 0 day 5 and day 14
  the blood tests were obtained to evaluate hematological counts (reticulocytes, hemoglobin, hematocrit, leukocytes), coagulation parameters (platelet count, partial thromboplastin and prothrombin times) and blood chemistry (glycemia, creatinine, urea, liver enzymes)
Change from Baseline Systolic Blood Pressure after each intervention | day 1-5
  The vital signs and the physical checkup was permanent before and after each application. The change of the baseline systolic blood pressure could be a criteria for suspension of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Amaro Gonzalez, PhD Eng, Principal Investigator — Centro Inmunologia Molecular CIM Havana Cuba; Teresita Rodríguez Obaya, PhD, Study Chair — Centro Immunologia Molecular CIM Havana Cuba; Iliana Sosa Teste, PhD, Principal Investigator — Centro Nacional Producción Animales de Laboratorio (CENPALAB) Cuba
Locations (2):
- Cuba (2):
  - Clinic of Movement Disorders, International Center for Neurological Restoration, Havana
  - Centro Inmunologia Molecular CIM, La Habana

REFERENCES:
- [Result] Pedroso I, Garcia M, Casabona E, Morales L, Bringas ML, Perez L, Rodriguez T, Sosa I, Ricardo Y, Padron A, Amaro D. Protective Activity of Erythropoyetine in the Cognition of Patients with Parkinson's Disease. Behav Sci (Basel). 2018 May 21;8(5):51. doi: 10.3390/bs8050051. eCollection 2018 May. PMID 29862060
- [Derived] Bringas Vega ML, Pedroso Ibanez I, Razzaq FA, Zhang M, Morales Chacon L, Ren P, Galan Garcia L, Gan P, Virues Alba T, Lopez Naranjo C, Jahanshahi M, Bosch-Bayard J, Valdes-Sosa PA. The Effect of Neuroepo on Cognition in Parkinson's Disease Patients Is Mediated by Electroencephalogram Source Activity. Front Neurosci. 2022 Jun 30;16:841428. doi: 10.3389/fnins.2022.841428. eCollection 2022. PMID 35844232
- [Derived] Garcia-Llano M, Pedroso-Ibanez I, Morales-Chacon L, Rodriguez-Obaya T, Perez-Ruiz L, Sosa-Teste I, Amaro-Gonzalez D, Bringas-Vega ML. Short-term Tolerance of Nasally-administered NeuroEPO in Patients with Parkinson Disease. MEDICC Rev. 2021 Jan;23(1):49-54. doi: 10.37757/MR2021.V23.N1.10. Epub 2021 Jan 30. PMID 33780423